CLINICAL TRIAL: NCT02927262
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the FLT3 Inhibitor Gilteritinib (ASP2215) Administered as Maintenance Therapy Following Induction/Consolidation Therapy for Subjects With FLT3/ITD AML in First Complete Remission
Brief Title: A Study of ASP2215 (Gilteritinib), Administered as Maintenance Therapy Following Induction/Consolidation Therapy for Subjects With FMS-like Tyrosine Kinase 3 (FLT3/ITD) Acute Myeloid Leukemia (AML) in First Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2215-CL-0302; 2016-001643-39 (EudraCT Number)
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Results first posted 2022-06-27 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia With FMS-like Tyrosine Kinase (FLT3) / Internal Tandem Duplication (ITD) Mutation
Keywords: Acute myeloid leukemia; First Complete Remission; gilteritinib; FLT3/ITD; AML; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gilteritinib (Experimental): Participants received gilteritinib 120 mg (three tablets of 40 mg) orally, once daily (QD) for up to 2 years or until a protocol-specified discontinuation criterion was met.
  Interventions: Drug: Gilteritinib
- Placebo (Placebo Comparator): Participants received gilteritinib matching placebo orally, QD for up to 2 years or until a protocol-specified discontinuation criterion was met.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gilteritinib — Oral tablet
  Other Names: ASP2215
  Arms: Gilteritinib
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study was to compare relapse-free survival (RFS) between participants with FMS-like tyrosine kinase 3 (FLT3) / internal tandem duplication (ITD) acute myeloid leukemia (AML) in first complete remission (CR1) and who were randomized to receive gilteritinib or placebo beginning after completion of induction/consolidation chemotherapy for a two-year period.

DETAILED DESCRIPTION:
Participants in CR1 were approached for this study after induction/consolidation therapy was complete and a decision not to proceed with transplantation was made or a suitable donor could not be identified. Participants were randomized in a 2:1 ratio to receive gilteritinib or placebo. Participants entered the screening period up to 14 days prior to the start of treatment. Participants were administered treatment over continuous 28-day cycles. Gilteritinib or placebo was given daily for up to 2 years. After treatment discontinuation, participants had a 30-day follow-up visit for safety, after which the participants entered the long-term follow up period for collection of subsequent AML treatment, remission status, and survival (cause of death and date of death). Final database lock will occur when last subject last follow-up visit is reached, per protocol. Study drug was not provided during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered an adult according to local regulation at the time of obtaining consent form (ICF).
* Subject consents to allow access to subject's diagnostic bone marrow aspirate or peripheral blood sample and/or the DNA derived from that sample, if available, that may be used to validate a companion diagnostic test for gilteritinib.
* Subject has confirmed morphologically documented AML, excluding acute promyelocytic leukemia (APL), in CR1 (including CRp and CRi). For the purposes of enrollment, CR will be defined as < 5% blasts in the bone marrow with no morphologic characteristics of acute leukemia (e.g., Auer rods) in the bone marrow with no evidence of extramedullary disease such as central nervous system involvement or granulocytic sarcoma.
* Subject will not proceed with transplantation as either a decision not to proceed with transplantation has been made either on the recommendation of the treating physician or by the patient or a suitable donor could not be identified.
* Subject is < 2 months from the start of the last cycle of consolidation and should have completed the recommended number of consolidations per local practice.
* Subject has had no use of investigational agents, with the exception of FLT3 inhibiting agents during induction and/or consolidation therapy, within the prior 4 weeks.
* Subject has had presence of the FLT3/ITD activating mutation in the bone marrow or peripheral blood as determined by the local institution at diagnosis.
* Subject has an ECOG performance status 0 to 2.
* Subject must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN), or if serum creatinine outside normal range, then glomerular filtration rate (GFR) > 40 mL/min/1.73m^2 as calculated with the 4-parameter Modification of Diet in Renal Disease (MDRD) equation.
  * Serum total bilirubin ≤ 2.5 mg/dL (43 μmol/L), except for subjects with Gilbert's syndrome.
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN.
  * Serum potassium and serum magnesium ≥ institutional lower limit of normal (LLN).
  * Absolute neutrophil count (ANC) ≥ 500/μl and platelets ≥ 20000/μl (unsupported by transfusions).
* Subject is suitable for oral administration of study drug.
* Female subject must either:

  * Be of nonchildbearing potential:
  * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
  * Documented surgically sterile or status posthysterectomy (at least 1 month prior to screening)
  * Or, if of childbearing potential,
  * Agree not to try to become pregnant during the study and for 6 months after the final study drug administration
  * And have a negative urine or serum pregnancy test at screening
  * And, if heterosexually active, agree to consistently use highly effective contraception per locally accepted standards (in addition to a barrier method) starting at screening and throughout the study period and for 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 2 months and 1 week after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Male subject and subject's female partners who are of childbearing potential must be using highly effective contraception per locally accepted standards (in addition to a barrier method) starting at screening and continue throughout the study period and for 4 months and 1 week after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 4 months and 1 week after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject has had prior allogeneic transplant.
* Subject has QTcF interval > 450 msec (average of triplicate determinations based on central reading).
* Subject with Long QT Syndrome.
* Subject with hypokalemia and hypomagnesemia at screening (defined as values below LLN).
* Subject has clinically active central nervous system leukemia.
* Subject is known to have human immunodeficiency virus infection.
* Subject has active hepatitis B or C.
* Subject has an uncontrolled infection. If a bacterial or viral infection is present, the subject must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to randomization. If a fungal infection is present, the subject must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to randomization.
* Subject has progressing infection defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Subject has uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, congestive heart failure New York Heart Association (NYHA) class 3 or 4 or subject has a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multigated acquisition (MUGA) scan performed within 1 month prior to study entry results in a left ventricular ejection fraction that is ≥ 45%.
* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP) 3A.
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P-glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5-hydroxytryptamine receptor 2B (5HT2BR) or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject has a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Subject has prior malignancies, except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.
* Subject has any condition which makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (73):
- United States (6):
  - Site US10017, Gainesville, Florida
  - Site US10030, Jacksonville, Florida
  - Site US10012, Chicago, Illinois
  - Site US10025, Syracuse, New York
  - Site US10007, Portland, Oregon
  - Site US10029, Greenville, South Carolina
- Site BR55002, Goiânia, Goiás, Brazil
- Canada (2):
  - Site CA15001, Halifax, Nova Scotia
  - Site CA15003, Toronto, Ontario
- Site CZ42001, Ostrava-Poruba, Czechia
- Site DK45002, Aarhus, Central Jutland, Denmark
- France (7):
  - Site FR33004, Brest, Finistere
  - Site FR33002, Tours, Indre-et-Loire
  - Site FR33014, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Site FR33007, Pierre-Bénite, Rhone
  - Site FR33001, Bayonne
  - Site FR33009, Mulhouse
  - Site FR33008, Nice
- Germany (2):
  - Site DE49001, Duisburg, North Rhine-Westphalia
  - Site DE49008, Stuttgart
- Greece (4):
  - Site GR30010, Athens, Attica
  - Site GR30004, Thessaloniki, Central Macedonia
  - Site GR30009, Athens
  - Site GR30007, Larissa
- Site HU36003, Nyíregyháza, Szabolcs-Szatmár-Bereg, Hungary
- Site IL97205, Jerusalem, Jerusalem, Israel
- Italy (6):
  - Site IT39011, Milan, Lombardy
  - Site IT39004, Castelfranco Veneto (TV), Treviso
  - Site IT39008, Bergamo
  - Site IT39005, Parma
  - Site IT39010, Reggio Emilia
  - Site IT39002, Roma
- Japan (12):
  - Site JP81018, Nagoya, Aichi-ken
  - Site JP81025, Matsuyama, Ehime
  - Site JP81002, Yoshida-gun, Fukui
  - Site JP81024, Sapporo, Hokkaido
  - Site JP81012, Kobe, Hyōgo
  - Site JP81004, Kanazawa, Ishikawa-ken
  - Site JP81009, Yokohama, Kanagawa
  - Site JP81014, Sendai, Miyagi
  - Site JP81023, Shimotsuke, Tochigi
  - Site JP81011, Tachikawa, Tokyo
  - Site JP81010, Aomori
  - Site JP81017, Okayama
- Poland (3):
  - Site PL48001, Olsztyn, Warmian-Masurian Voivodeship
  - Site PL48002, Bydgoszcz
  - Site PL48007, Poznan
- Portugal (2):
  - Site PT35106, Coimbra
  - Site PT35101, Porto
- Site RO40005, Bucharest, Romania
- Site RS38102, Belgrade, Serbia
- South Korea (8):
  - Site KR82005, Suwon, Gyeonggi-do
  - Site KR82014, Bucheon-si, Gyeonggido
  - Site KR82013, Goyang, Gyeonggido
  - Site KR82008, Namdong, Incheon Gwang'yeogsiv
  - Site KR82003, Hwasungun, Jeonranamdo
  - Site KR82012, Seoul, Seoul Teugbyeolsi
  - Site KR82006, Busan
  - Site KR82009, Seoul
- Site ES34009, Vitoria-Gasteiz, Alava, Spain
- Sweden (2):
  - Site SE46003, Stockholm, Stockholm County
  - Site SE46002, Lund
- Taiwan (3):
  - Site TW88605, Kaohsiung City
  - Site TW88604, Kaohsiung City
  - Site TW88603, Taipei
- United Kingdom (8):
  - Site GB44007, Exeter, Devon
  - Site GB44019, Plymouth, Devon
  - Site GB44006, Cottingham, East Riding Of Yorkshire
  - Site GB44018, London, London, City of
  - Site GB44002, Birmingham
  - Site GB44015, Cardiff
  - Site GB44020, Leeds
  - Site GB44004, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants diagnosed with FMS-like tyrosine kinase 3 (FLT3)/internal tandem duplication (ITD) acute myeloid leukemia (AML) in first complete remission (CR1), including complete remission with incomplete platelet recovery (CRp) and complete remission with incomplete hematologic recovery (CRi) for whom a decision not to proceed with transplantation was made, or a suitable donor could not be identified, were enrolled in this study.
Pre-assignment Details: Randomization was stratified based on:
  Age (<60 or ≥60 years), Geographic region (North America or Europe or rest of the world), Presence of Minimal Residual Disease (MRD) at screening (yes or no), Use of FLT3-inhibiting agents during induction/consolidation (yes or no).
Groups:
- Gilteritinib: Participants received gilteritinib 120 mg (three tablets of 40 mg) orally, QD for up to 2 years or until a protocol-defined discontinuation criterion was met.
- Placebo: Participants received gilteritinib matching placebo orally, QD for up to 2 years or until a protocol-defined discontinuation criterion was met.
Period: Treatment Period (Up to 744 Days)
Arm/Group | Gilteritinib | Placebo
Started | 63 | 35
Completed | 24 | 12
Not Completed | 39 | 23
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 1 | 0
Not completed — Treatment ended due to transplant procedure | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Becomes eligible for and proceeds to transplant | 0 | 1
Not completed — Participant relapsed and became eligible for and proceeded to transplant | 0 | 1
Not completed — Randomized in error | 1 | 0
Not completed — Participant was not eligible for the study | 1 | 0
Not completed — MRD positive | 0 | 1
Not completed — Disease Relapse | 23 | 18
Not completed — Adverse Event | 7 | 1
Not completed — Investigators decision to take participant off trial due to molecular relapse | 1 | 0
Not completed — Clinicians decision as suspected relapse | 0 | 1
Period: Long Term Follow-up (Up to 1201 Days)
Arm/Group | Gilteritinib | Placebo
Started | 60 (Participants who completed or discontinued treatment period were allowed to join the long term follow up period) | 35 (Participants who completed or discontinued treatment period were allowed to join the long term follow up period)
Did Not Enter Long Term Follow up Period | 3 | 0
Completed | 35 | 21
Not Completed | 25 | 14
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 23 | 12

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gilteritinib | Placebo | Total
Number analyzed (Participants) | 63 | 35 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (11.0) | 59.9 (13.9) | 60.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 51
  Male | 32 | 15 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 50 | 29 | 79
  Unknown or Not Reported | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 10 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 22 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 3 | 11
Age (<60 or ≥60 years) [Count of Participants; unit: Participants]
  <60 years | 24 | 13 | 37
  ≥60 years | 39 | 22 | 61
Geographic Region [Count of Participants; unit: Participants] — Geographical region was categorized as Europe, North America and Rest of the World.
  Participants
    North America | 5 | 4 | 9
    Europe | 40 | 20 | 60
    Rest of the world | 18 | 11 | 29
Presence of MRD [Count of Participants; unit: Participants] — Presence of MRD (yes/no) at screening per interatcive response technology (IRT) at randomization was reported. The presence of MRD will be "Yes" if log10-transformed overall FLT3/ITD mutation ratio was greater than -4
  Participants
    MRD = Yes | 8 | 6 | 14
    MRD = No | 55 | 29 | 84
Use of FLT3-inhibitors [Count of Participants; unit: Participants] — Use of FLT3 inhibitor (yes/no) during induction/consolidation per IRT at randomization was reported.
  Participants
    Use of FLT3 Inhibitor = Yes | 12 | 10 | 22
    Use of FLT3 Inhibitor = No | 51 | 25 | 76

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS) Per Independent Review Committee (IRC) Adjudication
Description: RFS was defined as the time from the date of randomization until the date of documented relapse or death from any cause, whichever occurred first. Relapse after complete remission (CR) [including complete remission with incomplete platelet recovery (CRp) and Complete remission with incomplete hematologic recovery (CRi)], was defined as bone marrow blasts 5% or higher (not attributable to regenerating bone marrow), any circulating blasts, any extra-medullary blast foci as per Revised International Working Group (IWG) criteria.
  Participants were classified as:
  CRi, if they fulfilled all the criteria for CR except for incomplete hematological recovery with residual neutropenia < 1 × 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence was not required.
  CRp, if they achieved CR except for incomplete platelet recovery (< 100 × 10^9/L).
  RFS was estimated using Kaplan-Meier estimates. hazard ratio (HR), cox proportional hazards model (CHM)
Time Frame: From the date of randomization until the date of documented relapse, or death; (Median time on study drug was 427 days for gilteritinib group and 212 days for placebo group)
Population: The full analysis set (FAS) consisted of all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 63 | 35
Months | 24.02 [14.06 to NA] — Upper limit was not estimable due to low number of events | 15.84 [3.02 to NA] — Upper limit was not estimable due to low number of events
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Test type: Superiority; p = 0.163, Log Rank; Hazard Ratio (HR) = 0.738, 95% CI 2-sided [0.407 to 1.336] — HR & 95% CI are based on CHM. Assuming proportional hazards, HR < 1 indicates a reduction in hazard rate in favor of gilteritinib arm. Stratification factors:age, geographic region, presence of MRD at screening, use of FLT3 inhibiting agents per IRT

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. OS was estimated using Kaplan-Meiers method.
Time Frame: From the date of randomization until the date of death from any cause; (Median time on study drug was 427 days for gilteritinib group and 212 days for placebo group)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 63 | 35
Months | NA [30.42 to NA] — Median and upper limit were not estimable due to low number of events | NA [43.56 to NA] — Median and upper limit were not estimable due to low number of events
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Test type: Superiority; p = 0.627, Log Rank; Hazard Ratio (HR) = 1.130, 95% CI [0.540 to 2.364] — HR & 95%CI are based on CHM. Assuming proportional hazards, HR < 1 indicates a reduction in hazard rate in favor of gilteritinib arm. Stratification factors: age, geographic region, presence of MRD at screening, use of FLT3 inhibiting agents per IRT

3. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from the date of randomization until the date of documented relapse or discontinuation of the treatment, or initiation of other anti-leukemic treatment or death from any cause, whichever occurred first. Relapse after CR (including CRp and CRi), was defined as bone marrow blasts 5% or higher (not attributable to regenerating bone marrow), any circulating blasts, any extra-medullary blast foci as per Revised IWG criteria.
  Participants were classified as:
  CRi, if they fulfilled all the criteria for CR except for incomplete hematological recovery with residual neutropenia < 1 × 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence was not required.
  CRp, if they achieved CR except for incomplete platelet recovery (< 100 × 10^9/L).
  EFS was estimated using Kaplan-Meier's method.
Time Frame: From date of randomization until the date of documented relapse or discontinuation of the treatment, or initiation of other anti-leukemic treatment or death from any cause; (Median time on study drug was 427 days for gilteritinib and 212 days for Placebo)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 63 | 35
Months | 14.06 [9.89 to 23.72] | 6.74 [2.86 to 21.95]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Test type: Superiority; p = 0.296, Log Rank; Hazard Ratio (HR) = 0.862, 95% CI 2-sided [0.510 to 1.455] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Quantitative Minimal Residual Disease Measured as Log10-transformed Overall FLT3/ITD Mutation Ratio at Months 3, 6, 12, 24/End of Treatment (EoT)
Description: MRD was measured from bone marrow samples. FLT3/ITD mutation ratio was measured in relation to total FLT3. For a participant with multiple ITD mutations, the overall FLT3/ITD mutation ratio was calculated from the sum of all ITD mutations. Absence of Minimal Residual Disease (MRD) is defined as log10-transformed overall FLT3/ITD mutation ratio ≤ -4.
Time Frame: Baseline and months 3, 6, 12, 24/EoT
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 48 | 22
Ratio
  Month 3 | 0.14 (0.96) | 0.14 (1.46)
  Month 6: number analyzed (Participants) | 44 | 17
  Month 6 | 0.07 (0.92) | -0.17 (0.79)
  Month 12: number analyzed (Participants) | 32 | 14
  Month 12 | -0.11 (0.60) | -0.34 (0.67)
  Month 24/EoT: number analyzed (Participants) | 28 | 14
  Month 24/EoT | -0.12 (1.08) | 0.23 (1.63)
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Month 3; Test type: Superiority; p = 0.970, ANCOVA — 2-sided P-value from analysis of covariance (ANCOVA) including treatment, age group, geographic region and use of FLT3-inhibiting agents per IRT as fixed factors and baseline score as covariate
Statistical Analysis 2: Comparison: Gilteritinib vs Placebo; Month 6; Test type: Superiority; p = 0.415, ANCOVA — 2-sided P-value from ANCOVA including treatment, age group, geographic region and use of FLT3-inhibiting agents per IRT as fixed factors and baseline score as covariate
Statistical Analysis 3: Comparison: Gilteritinib vs Placebo; Month 12; Test type: Superiority; p = 0.271, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Gilteritinib vs Placebo; Month 24/EoT; Test type: Superiority; p = 0.179, ANCOVA — [p-value comment as in outcome 4, analysis 2]

5. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a participant administered a study drug, which does not necessarily have to have a causal relationship with treatment. It can, be any unfavorable and unintended sign, symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product whether considered related to the medicinal product. An AE is considered "serious" if, it results in results in death, is life-threatening (an AE is considered "life-threatening" if, its occurrence places the participant at immediate risk of death, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, Requires inpatient hospitalization (except for planned procedures as allowed per study) or leads to prolongation of hospitalization.
  TEAE was defined as an AE observed after starting administration of the study drug through 30 days after the last dose.
Time Frame: From first dose date up to 30 days after last dose or data cut-off date 25-May 2021 (Maximum treatment duration was 744 days)
Population: The safety analysis set (SAF) consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 62 | 35
Participants
  TEAE | 58 | 33
  Drug-Related TEAE | 51 | 20
  TEAE before Relapse | 57 | 28
  Drug-Related TEAE before Relapse | 51 | 15
  Serious TEAE | 24 | 14
  Drug-Related Serious TEAE | 10 | 3
  TEAE Leading to Death | 1 | 1
  Drug-Related TEAE Leading to Death | 0 | 1
  TEAE Leading to Withdrawal of Treatment | 15 | 6
  Drug-Related TEAE Leading to Withdrawal of Treatment | 5 | 2
  TEAE Leading to Dose Reduction | 15 | 1
  Drug-Related TEAE Leading to Dose Reduction | 14 | 1
  TEAE Leading to Dose Interruption | 35 | 4
  Drug-Related TEAE Leading to Dose Interruption | 31 | 1
  Grade 3 or Higher Treatment-Emergent Adverse Events | 42 | 18
  Grade 3 or Higher Drug-related TEAE | 33 | 4
  Death | 20 | 11

6. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score
Description: ECOG performance status was measured on an 6 point scale. 0-Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
  Number of participants with ECOG PS was reported. ECOG PS grades with zero participants were not reported.
Time Frame: Months 1, 2, 3, 4, 5, 6, 8, 10. 12, 14, 16, 18, 20, 22 and 24/EoT
Population: Safety population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 62 | 35
Participants
  Baseline: Grade 0 | 39 | 22
  Baseline: Grade 1 | 23 | 13
  Month 2: Grade 0: number analyzed (Participants) | 54 | 28
  Month 2: Grade 0 | 38 | 18
  Month 2: Grade 1: number analyzed (Participants) | 54 | 28
  Month 2: Grade 1 | 16 | 9
  Month 2: Grade 2: number analyzed (Participants) | 54 | 28
  Month 2: Grade 2 | 0 | 1
  Month 3: Grade 0: number analyzed (Participants) | 52 | 25
  Month 3: Grade 0 | 33 | 20
  Month 3: Grade 1: number analyzed (Participants) | 52 | 25
  Month 3: Grade 1 | 19 | 4
  Month 3: Grade 2: number analyzed (Participants) | 52 | 25
  Month 3: Grade 2 | 0 | 1
  Month 4: Grade 0: number analyzed (Participants) | 49 | 22
  Month 4: Grade 0 | 37 | 16
  Month 4: Grade 1: number analyzed (Participants) | 49 | 22
  Month 4: Grade 1 | 12 | 6
  Month 5: Grade 0: number analyzed (Participants) | 46 | 21
  Month 5: Grade 0 | 35 | 17
  Month 5: Grade 1: number analyzed (Participants) | 46 | 21
  Month 5: Grade 1 | 11 | 4
  Month 6: Grade 0: number analyzed (Participants) | 43 | 19
  Month 6: Grade 0 | 32 | 17
  Month 6: Grade 1: number analyzed (Participants) | 43 | 19
  Month 6: Grade 1 | 11 | 2
  Month 8: Grade 0: number analyzed (Participants) | 41 | 18
  Month 8: Grade 0 | 32 | 12
  Month 8: Grade 1: number analyzed (Participants) | 41 | 18
  Month 8: Grade 1 | 8 | 6
  Month 8: Grade 2: number analyzed (Participants) | 41 | 18
  Month 8: Grade 2 | 1 | 0
  Month 10: Grade 0: number analyzed (Participants) | 37 | 17
  Month 10: Grade 0 | 29 | 14
  Month 10: Grade 1: number analyzed (Participants) | 37 | 17
  Month 10: Grade 1 | 8 | 3
  Month 12: Grade 0: number analyzed (Participants) | 35 | 17
  Month 12: Grade 0 | 24 | 14
  Month 12: Grade 1: number analyzed (Participants) | 35 | 17
  Month 12: Grade 1 | 11 | 3
  Month 14: Grade 0: number analyzed (Participants) | 30 | 16
  Month 14: Grade 0 | 21 | 13
  Month 14: Grade 1: number analyzed (Participants) | 30 | 16
  Month 14: Grade 1 | 9 | 3
  Month 16: Grade 0: number analyzed (Participants) | 28 | 13
  Month 16: Grade 0 | 22 | 11
  Month 16: Grade 1: number analyzed (Participants) | 28 | 13
  Month 16: Grade 1 | 4 | 2
  Month 16: Grade 2: number analyzed (Participants) | 28 | 13
  Month 16: Grade 2 | 2 | 0
  Month 18: Grade 0: number analyzed (Participants) | 27 | 14
  Month 18: Grade 0 | 19 | 13
  Month 18: Grade 1: number analyzed (Participants) | 27 | 14
  Month 18: Grade 1 | 8 | 1
  Month 20: Grade 0: number analyzed (Participants) | 25 | 14
  Month 20: Grade 0 | 18 | 13
  Month 20: Grade 1: number analyzed (Participants) | 25 | 14
  Month 20: Grade 1 | 7 | 1
  Month 22: Grade 0: number analyzed (Participants) | 24 | 13
  Month 22: Grade 0 | 20 | 11
  Month 22: Grade 1: number analyzed (Participants) | 24 | 13
  Month 22: Grade 1 | 4 | 2
  Month 24/EoT: Grade 0: number analyzed (Participants) | 51 | 28
  Month 24/EoT: Grade 0 | 34 | 20
  Month 24/EoT: Grade 1: number analyzed (Participants) | 51 | 28
  Month 24/EoT: Grade 1 | 14 | 6
  Month 24/EoT: Grade 2: number analyzed (Participants) | 51 | 28
  Month 24/EoT: Grade 2 | 1 | 0
  Month 24/EoT: Grade 3: number analyzed (Participants) | 51 | 28
  Month 24/EoT: Grade 3 | 1 | 1
  Month 24/EoT: Grade 4: number analyzed (Participants) | 51 | 28
  Month 24/EoT: Grade 4 | 1 | 1

ADVERSE EVENTS:
Time Frame: From the date of randomization up to end of study (85 months and 9 days)
Description: All randomized participants for All-cause mortality. Safety Population (SAF) for serious adverse events and non-serious adverse events. The SAF consisted of all randomized participants who took at least 1 dose of study intervention and was used for safety analyses.
Arm/Group | Gilteritinib | Placebo
All-Cause Mortality (participants affected / at risk) | 24/63 | 12/35
Serious Adverse Events (participants affected / at risk) | 24/62 | 14/35
Other Adverse Events (participants affected / at risk) | 53/62 | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=62) | Placebo (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Systemic mastocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (2) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=62) | Placebo (N=35)
Anaemia (Blood and lymphatic system disorders) | 5 (8) | 5 (8)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (32) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (17) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Dry eye (Eye disorders) | 5 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (3)
Nausea (Gastrointestinal disorders) | 8 (10) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Fatigue (General disorders) | 10 (10) | 3 (4)
Malaise (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 3 (3) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 3 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (5) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (11) | 6 (11)
Otitis media (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3)
Urinary tract infection (Infections and infestations) | 3 (7) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 8 (17) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 7 (12) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (6)
Blood creatine phosphokinase increased (Investigations) | 18 (37) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 7 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 12 (46) | 3 (5)
Platelet count decreased (Investigations) | 12 (24) | 4 (10)
Weight increased (Investigations) | 8 (11) | 2 (4)
White blood cell count decreased (Investigations) | 6 (24) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (7) | 2 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9) | 4 (4)
Headache (Nervous system disorders) | 5 (9) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (5) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02927262/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02927262/SAP_001.pdf